CLINICAL TRIAL: NCT03681275
Title: A Clinical Trial of JAK Inhibition to Prevent Ventilator-induced Diaphragm Dysfunction
Brief Title: Janus Kinase Inhibition to Prevent Ventilator-induced Diaphragm Dysfunction
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Joseph B. Shrager, MD, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB-47826; 3R01AG069858-02W1 (NIH)
Record Dates: First submitted 2018-09-20; First posted 2018-09-24 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Diaphragm Injury
Keywords: Ventilator-induced Diaphragm Dysfunction
MeSH Terms: interventions — tofacitinib

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tofacitinib (Experimental): Patient will receive two days treatment with tofacitinib prior to the surgery.
  Interventions: Drug: Tofacitinib 10 MG [Xeljanz]
- Placebo (Placebo Comparator): Patient will receive two days treatment with placebo prior to the surgery.
  Interventions: Drug: Placebo to match Tofacitinib

INTERVENTIONS:
Drug: Tofacitinib 10 MG [Xeljanz] — administered twice daily for two days
  Other Names: XELJANZ
  Arms: Tofacitinib
Drug: Placebo to match Tofacitinib — administered twice daily for two days
  Arms: Placebo

SUMMARY:
We intend, with this study, to prove that blocking the molecular mechanisms whose blockade prevents VIDD in animals, will indeed prevent the development of VIDD in humans as well. We believe that this evidence will serve as the required basis for proceeding with large, ICU-based clinical trial(s) of a drug to prevent VIDD.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing esophagectomy

Exclusion Criteria:

* Patients with more than mild pulmonary dysfunction
* Patients with any neuromuscular disease that might compromise diaphragm function
* Patients with abnormal liver or kidney function
* Patients taking any immunosuppressant medication (including prednisone) or antifungal medications
* History of tuberculosis
* Weight loss of >5% of body weight over previous 6 months
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-09-03 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Prevention of ventilator-induced diaphragm dysfunction by JAK inhibition | 5-6 years
  Change in the force deficit that develops between the first and second muscle biopsies in the drug-treated vs. placebo groups

SECONDARY OUTCOMES:
Increase in muscle strength due to JAK inhibition | 4-5 years
  Difference in force generated by muscle biopsies taken at time point 1 (pre-mechanical ventilation) from the drug-treated vs placebo groups

OTHER OUTCOMES:
Exploratory: Determine mechanisms of changes in muscle strength and ventilator-induced diaphragm dysfunction by JAK inhibition. | 4-6 years
  Compare differences in muscle between the drug-treated and placebo groups in mitochondrial function and oxidative stress (ATP levels, citrate synthase activity, succinate dehydrogenase activity, mitochondrial respiration rate, activity of mitochondial enzymatic compexes).
Exploratory: Determine mechanisms of changes in muscle strength and ventilator-induced diaphragm dysfunction by JAK inhibition. | 4-6 years
  Compare differences in muscle between the drug-treated and placebo groups in proteolytic pathways (quantitative PCR for atrogein, MuRF1, and FoxO gene expression, western blot analysis for protein levels of these and protein polyubiquitination, proteasomal activity, qPCR and western blots for expression of LC3).
Exploratory: Determine mechanisms of changes in muscle strength and ventilator-induced diaphragm dysfunction by JAK inhibition. | 4-6 years
  Compare differences in muscle between the drug-treated and placebo groups in transcriptomic gene profiling, and metabolomic profiling..

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Shrager, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Medical Center, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD.

REFERENCES:
- [Background] Shrager JB, Wang Y, Lee M, Nesbit S, Trope W, Konsker H, Fatodu E, Berry MS, Poulstides G, Norton J, Burdon T, Backhus L, Cooke R, Tang H. Rationale and design of a mechanistic clinical trial of JAK inhibition to prevent ventilator-induced diaphragm dysfunction. Respir Med. 2021 Nov-Dec;189:106620. doi: 10.1016/j.rmed.2021.106620. Epub 2021 Sep 21. PMID 34655959
- [Background] Shrager JB, Randle R, Lee M, Ahmed SS, Trope W, Lui N, Poultsides G, Liou D, Visser B, Norton JA, Nesbit SM, He H, Kapula N, Wallen B, Fatodu E, Sadeghi CA, Konsker HB, Elliott I, Guenthart B, Backhus L, Cooke R, Berry M, Tang H. JAK inhibition with tofacitinib rapidly increases contractile force in human skeletal muscle. Life Sci Alliance. 2024 Aug 9;7(11):e202402885. doi: 10.26508/lsa.202402885. Print 2024 Nov. PMID 39122555